CLINICAL TRIAL: NCT06103656
Title: Double-Blind, Placebo-Controlled Phase 2 Study to Assess Safety and Efficacy of Chinese Herbal Therapy and Multiple Food Allergen Oral Immunotherapy
Brief Title: E-B-FAHF-2, Multi OIT and Xolair for Food Allergy
Acronym: FAHF-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02879006
Record Dates: First submitted 2023-09-20; First posted 2023-10-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator::Chinese Herbal Medication (Experimental): Interventions:
  - Drug: Chinese Herbal Medication (E-B-FAHF-2), dose level was determined using the subject's weight at the screening visit (>20-30 kg = 5 capsules daily, >30-70 kg = 8 capsules daily, and >70 kg = 10 capsules daily)
  Interventions: Drug: Drug: Chinese Herbal Medication; Drug: Drug: Omalizumab
- Placebo Comparator: Placebo (Placebo Comparator): Interventions:
  * Drug: Placebo. Placebo capsules were identical in appearance but contained corn starch
  * Drug: Omalizumab. Omalizumab was dosed as per the product insert
  * Drug: Multi OIT. An initial rush dose to a maximum of 250 mg of protein of each allergen (total 270 mg of protein) and up-dosing every 2 weeks until the maintenance dose of 1000mg was reached.
  Interventions: Drug: Drug: Placebo

INTERVENTIONS:
Drug: Drug: Chinese Herbal Medication — Capsules, 26 month course, starting 2 months pre-OIT.
  Other Names: E-B-FAFH-2
  Arms: Active Comparator::Chinese Herbal Medication
Drug: Drug: Placebo — Placebo capsules that look identical to E-B-FAHF-2 containing corn starch, 26 month course, starting 2 months pre-OIT
  Other Names: Placebo Chinese Herb
  Arms: Placebo Comparator: Placebo
Drug: Drug: Omalizumab — 4 months course, starting 2 months pre-OIT through the 2 month build-up phase
  Other Names: Xolair®
  Arms: Active Comparator::Chinese Herbal Medication

SUMMARY:
The purpose of this study is testing the use of Enhanced-Butanol purified-Food Allergy Herbal Formula-2 (E-B-FAHF-2) Chinese herbal therapy in combination with multi-food oral immunotherapy (OIT) and Xolair® (Omalizumab) to help children and adults who are allergic to foods be able to safely tolerate food allergens. Specifically in this protocol, the food allergens are milk, egg, peanut, almond, cashew, hazelnut, walnut, sesame, and/or wheat. Omalizumab is considered an investigational drug for the treatment of food allergies in children and adults. Investigational means it has not been approved by the Food and Drug Administration (FDA) for use in the U.S. The researchers hope to learn whether the addition of Chinese herbal therapy (E-B-FAHF-2) can improve the outcome of sustained unresponsiveness (which is the ability to consume a food allergen and pass an oral food challenge after being off treatment for 3 months) as compared to placebo (i.e. subjects with OIT/Omalizumab + herbal vs. OIT/Omalizumab + placebo), and will help adults and children be able to safely ingest the foods they are allergic to.

DETAILED DESCRIPTION:
Prior studies have shown that this Chinese herbal formulation is safe and well-tolerated in food allergic individuals. While oral immunotherapy (OIT) can lead to desensitization, it remains uncertain whether this treatment can lead to lasting protection. Therefore, this study aims to use the Chinese herbal formula in combination with OIT to determine whether sustained protection can be achieved. All subjects will receive multi-allergen OIT, along with a 4 month course of omalizumab to provide added safety for the initial dose escalation and build up phases. Subjects will be randomized to receive active Chinese herbal formula or placebo. Subjects will be treated with OIT for 2 years and then food challenges will be performed to assess for desensitization. For those who achieve desensitization, all treatments will be discontinued and food challenges will be performed 3 months later to assess for sustained unresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* 6 through 40 years
* At least one of the following for each of the 3 study allergens: serum immunoglobulin E (IgE) >4000 U/L or skin -prick test >6mm
* dose limiting symptoms at a cumulative dose of <=444 mg protein for 3 allergens as screening double-blind, placebo-controlled food challenge
* use of an effective method of contraception by females of child-bearing potential
* ability to ingest oat or corn with no allergic reaction

Exclusion Criteria:

* If baked milk or egg are tolerated (assessed by clinical report), then milk or egg may not be included as a study allergen
* Any disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, and serious ventricular arrhythmias
* History of other chronic disease requiring therapy (other than asthma, atopic dermatitis, or rhinitis)
* History of eosinophilic gastrointestinal disease
* Current participation in any other interventional study
* Investigational drug use within 90 days
* Subject is on build-up phase of any allergen immunotherapy (prior to maintenance dosing)
* Current uncontrolled moderate to severe asthma as defined by:
* Forced Expiratory Volume-1 (FEV1) value <80% predicted or any clinical features of moderate or severe persistent asthma baseline severity (as defined by the 2007 NHLBI Guidelines) and greater than high daily doses of inhaled corticosteroids (as defined for children and adults using dosing tables from the 2007 NHLBI Guidelines).
* Use of steroid medications in the following manners: history of daily oral steroid dosing for >1 month during the past year, having 1 burst or steroid course within the past 6 months, or having >1 burst oral steroid course within the past 12 months.
* Asthma requiring >1 hospitalization in the past year for asthma or >1 Emergency Department (ED) visit in the past 6 months for asthma.
* Use of systemic steroid medications (Intravenous, Intramuscular or oral) for indications other than asthma for > 3 weeks within the past 6 months
* Inability to discontinue antihistamines for the initial day of escalation, skin testing or DBPCFC
* Use of Xolair® (omalizumab) within the past 6 months
* Known sensitivity to Xolair® (omalizumab) or to the class of study drugs
* Body weight more than 90 kg, or subjects with weight-IgE combination that yields a dose requirement greater than 600 mg dosing
* Use of beta-blockers (oral), Angiotensinogen converting enzyme (ACE) inhibitors, angiotensin-receptor blockers or calcium channel blockers
* Pregnancy or lactation
* Inability to swallow placebo capsules
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Sustained unresponsiveness to cumulative dose of 4,444 mg protein | 29 months
  Sustained unresponsiveness evaluated by the absence of dose-limiting symptoms to a cumulative dose of 4,444 mg protein.

SECONDARY OUTCOMES:
Desensitization to 4444mg protein | 26 months
  Number of participants in the E-B-FAFH-2 group (EOIT) tolerating a cumulative dose of 4,4444mg of food allergen protein.
High level desensitization to 7444mg protein or higher | 26 months
  Number of participants tolerating a cumulative dose of 7,444mg or higher (max of 10,444mg) to food allergen protein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang J, Wood RA, Raymond S, Suarez-Farinas M, Yang N, Sicherer SH, Sampson HA, Li XM. Double-Blind, Placebo-Controlled Study of E-B-FAHF-2 in Combination With Omalizumab-Facilitated Multiallergen Oral Immunotherapy. J Allergy Clin Immunol Pract. 2023 Jul;11(7):2208-2216.e1. doi: 10.1016/j.jaip.2023.03.051. Epub 2023 Apr 20. PMID 37087097